CLINICAL TRIAL: NCT00194116
Title: Double-blind, Placebo-Controlled Divalproex Sodium ER in Bipolar I or Bipolar II Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Keming Gao, Director, Mood and Anxiety Clinic, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHHS 08-03-07
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Divalproex Sodium ER (Experimental)
  Interventions: Drug: Divalproex Sodium ER
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Divalproex Sodium ER — Tablets will be available in 250mg and 500mg strengths. Divalproex will be titrated to a minimum blood level of 50 mg/L. However, the investigators will titrate divalproex to the maximum tolerable dose with an expected average dose of 2000mg per day. By dosing in this manner, all subjects will have a minimum blood level of 50 mg/L, but the mean level is likely to be considerably higher.
  Other Names: Depakote ER
  Arms: Divalproex Sodium ER
Drug: Placebo — . Tablets will be available in 250mg and 500mg strengths. Divalproex will be titrated to a minimum blood level of 50 mg/L. However, the investigators will titrate divalproex to the maximum tolerable dose with an expected average dose of 2000mg per day. By dosing in this manner, all subjects will have a minimum blood level of 50 mg/L, but the mean level is likely to be considerably higher.
  Arms: Placebo

SUMMARY:
Double-Blind, Placebo-Controlled Divalproex Sodium ER in Bipolar I or Bipolar II Depression Previously Diagnosed and Treated as Recurrent Major Depression: This study recruits males and females aged 18 - 70 who currently meet diagnostic criteria for bipolar I or bipolar II disorder and are currently experiencing an episode of major depression. Patients are randomized to double-blind treatment with divalproex sodium ER or placebo and remain in the study for up to six weeks. This six-week double-blind treatment period is followed by an open-label treatment period of six months duration. This study is sponsored by Abbott Laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Subject must give consent to participate in the study and sign and date the IRB approved written informed consent form prior to the initiation of any study procedures
* Subject must be between the ages of 18 and 70
* Subject must have a diagnosis of bipolar I or II.
* Subject must be currently depressed as confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* Subject must have a baseline Montgomery-Asberg Depression Scale (MADRS) score of >19 and Young Mania Rating Scale (YMRS) score of <12
* Women of childbearing potential must be nonpregnant/nonlactating and using adequate contraception if sexually active
* Subject must not be using any concomitant psychotropic medications during the acute phase except prn benzodiazepines

Exclusion Criteria:

* Subjects lacks the capacity to provide informed consent
* Subject has currently or previously used divalproex or Dvpx-ER
* Subject is a serious suicide risk or has medically unstable conditions as judged by the investigators
* Subject has any alcohol, cocaine, or cannabis dependence within 3 months of study entry
* Subject has any cocaine, hallucinogens, opiates, crystal methamphetamine, or MMDA abuse within 3 months of study entry

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — Case Western Reserve University / University Hospitals of Cleveland
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Muzina DJ, Gao K, Kemp DE, Khalife S, Ganocy SJ, Chan PK, Serrano MB, Conroy CM, Calabrese JR. Acute efficacy of divalproex sodium versus placebo in mood stabilizer-naive bipolar I or II depression: a double-blind, randomized, placebo-controlled trial. J Clin Psychiatry. 2011 Jun;72(6):813-9. doi: 10.4088/JCP.09m05570gre. Epub 2010 Aug 24. PMID 20816041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Divalproex Sodium ER | Placebo
Started | 26 | 28
Completed | 13 | 13
Not Completed | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Divalproex Sodium ER | Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (10.3) | 38.8 (14.4) | 39.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
DSM-IV Diagnosis [Count of Participants; unit: Participants]
  Bipolar I Disorder | 10 | 10 | 20
  Bipolar II Disorder | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS total scores range from 0-60, where higher scores are indicative of more depression.
Time Frame: Acute phase (week0-week6)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale | -9.64 (1.49) | -5.32 (1.40)

2. Secondary Outcome: Change in Young Mania Rating Scale (YMRS) Total Score
Description: YMRS Scores range from 0 to 60 where higher scores are indicative of more mania.
Time Frame: Acute phase (week0-week6)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale | -0.54 (5.04) | -0.46 (3.28)

3. Secondary Outcome: Change in General Behavior Inventory (GBI) Depression Scale Score
Description: GBI Depression Scale Scores range from 46-184, where higher scores are indicative of more depression.
Time Frame: Acute phase (week0-week6)
Population: Not all subjects completed the GBI at study end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -11.56 (14.0) | 0.9 (18.4)

4. Secondary Outcome: Change in General Behavior Inventory (GBI) Hypomanic/Biphasic Scale Score
Description: GBI Hypomanic/Biphasic Scale scores range from 28-112, where higher scores are indicative of more hypomanic/manic symptoms.
Time Frame: Acute phase (week0-week6)
Population: Not all subjects completed the GBI at study end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -7.2 (8.3) | -6.8 (7.3)

5. Secondary Outcome: Change in Short Form Health Survey (SF-36) Physical Component Summary Score
Description: SF-36 Physical Component Summary scores range from 0-100, with a higher score indicating better physical health.
Time Frame: Acute phase (week0-week6)
Population: Not all subjects completed the SF-36 at study end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 18 | 14
units on a scale | -3.4 (15.7) | -4.2 (9.2)

6. Secondary Outcome: Change in Short Form Health Survey (SF-36) Mental Component Summary Score
Description: SF-36 Mental Component Summary scores range from 0-100, with a higher score indicating better mental health.
Time Frame: Acute phase (week0-week6)
Population: Not all subjects completed the SF-36 at study end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 18 | 14
units on a scale | 17.9 (18.4) | 13.5 (15.7)

7. Secondary Outcome: Change in Hamilton Anxiety Rating Scale (HAMA) Total Score
Description: HAMA Scores range from 0 to 56 where higher scores are indicative of more anxiety.
Time Frame: Acute phase (week0-week6)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Divalproex Sodium ER | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale | -4.6 (4.6) | -3.5 (7.0)

ADVERSE EVENTS:
Arm/Group | Divalproex Sodium ER | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 13/26 | 5/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Divalproex Sodium ER (N=26) | Placebo (N=28)
Nausea (Gastrointestinal disorders) | 9 (26) | 4 (28)
Increased Appetite (General disorders) | 4 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (3)
Dry Mouth (General disorders) | 3 (3) | 1 (1)
Stomach Cramps (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No